CLINICAL TRIAL: NCT06778616
Title: Frequency and Predictors of Recurrent Spontaneous Bacterial Peritonitis in Cirrhotic Patients in Al Rajhi University Hospital
Brief Title: Frequency and Predictors of Recurrent SBP in Cirrhotic Patients in Al Rajhi University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Moussa Hussein Hassan, Principal Investigator, Assiut University
Other Study IDs: Recurrence of SBP
Record Dates: First submitted 2024-09-09; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Spontaneous Bacterial Peritonitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
* Assess the frequency of recurrent SBP in ascitic cirrhotic patients.
* Determine the predictive factors of recurrence after the first episode of SBP in ascitic cirrhotic patients

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis (SBP) is a common complication in cirrhotic patients. The prevalence of SBP in hospitalized patients and the mortality rate were reported to be 10%-30% and 30%-50%, respectively.

SBP has been considered a life-threatening infection that requires a prompt diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Any cirrhotic patient above the age of 18 years old of both sexes, having a first episode of SBP will be included in our study.

  1. The diagnosis of cirrhosis was based on clinical manifestation (ascites, splenomegaly, lower limb edema and/or esophageal varices by upper gastrointestinal endoscopy), laboratory findings and radiological (abdominal ultrasonography), or liver histology.
  2. The diagnosis of SBP was based on a neutrophil cell count of 250 cell or more per mm3 with or without culture positivity of ascitic fluid, in the absence of hemorrhagic ascites and secondary peritonitis.

Exclusion Criteria:

* Any patient with one or more of the following criteria will be excluded:

  1. Patients with bacterial ascites defined by a positive culture of ascitic fluid associated with a neutrophil cell count less than 250 cell per mm3 in the ascitic fluid.
  2. Patients presenting with empyema or bacterial peritonitis secondary to an intra-abdominal organ perforation or surgical operation

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any cirrhotic patient above the age of 18 years old of both sexes, having a first episode of SBP will be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and Predictors of Recurrent Spontaneous Bacterial Peritonitis in Cirrhotic Patients in Al Rajhi University Hospital. | One year
  Determine the frequency of recurrent SBP after its management within one year

SECONDARY OUTCOMES:
Predictors of recurrent SBP | One year
  Determining risk factors of recurrent SBP

CONTACTS AND LOCATIONS:
Overall Officials: Marwa A Ahmed, MD, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assiut Faculty of Medicine, Asyut, Asyut Governorate
  - Assiut University, Asyut, Asyut Governorate

REFERENCES:
- [Background] Moalla M, Elleuch N, Dahmani W, Hammami A, Ameur WB, Slama AB, Brahem A, Ajmi S, Ksiaa M, Jaziri H, Jmaa A. Predictive factors of recurrence in spontaneous bacterial peritonitis in Tunisian patients with cirrhosis. Future Sci OA. 2023 Apr 17;9(5):FSO857. doi: 10.2144/fsoa-2023-0016. eCollection 2023 Jun. PMID 37180608